CLINICAL TRIAL: NCT02576444
Title: A Phase II Study of the PARP Inhibitor Olaparib (AZD2281) Alone and in Combination With AZD1775, AZD5363, or AZD6738 in Advanced Solid Tumors
Brief Title: OLAParib COmbinations
Acronym: OLAPCO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was paused during COVID and without the ability to initiate the 4th arm in the study, the decision was to terminate the study in 2022.
Sponsor: Joseph Paul Eder (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Vanderbilt-Ingram Cancer Center (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Joseph Paul Eder, Professor of Medicine; Clinical Director, Early Drug Development Program, Yale University
Organization: Yale University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1508016363
Record Dates: First submitted 2015-10-12; First posted 2015-10-15 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — olaparib; capivasertib; adavosertib; ceralasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): Patients with cholangiocarcinoma harboring IDH 1/2 tumors will be treated with olaparib. Patients with tumors harboring mutation in HDR genes will be treated with olaparib.
  Interventions: Drug: AZD2281
- Group 2 (Experimental): Patients with tumors harboring PTEN, PIK3CA, AKT, or ARID1A mutations or other molecular aberrations leading to dysregulation of the PI3K/AKT pathway will be treated with AZD5363 plus olaparib.
  Interventions: Drug: AZD2281; Drug: AZD5363
- Group 3 (Experimental): Patients with tumors harboring either TP53 or KRAS mutations or mutations in KRAS and TP53 will be treated with AZD1775 plus olaparib. TP53 mutations must be found on the TP53 mutation eligibility list.
  Interventions: Drug: AZD2281; Drug: AZD1775
- Group 4 (Experimental): Patients with tumors harboring mutations in HDR genes, including ATM, CHK2, APOBEC, MRE11 complex, will be treated with AZD6738 and olaparib.
  Interventions: Drug: AZD2281; Drug: AZD6738

INTERVENTIONS:
Drug: AZD2281 — Patients will be administered olaparib orally twice daily (bid) at 300 mg. Two (2) x 150 mg olaparib tablets should be taken at the same times each morning and evening of each day, approximately 12 hours apart with approximately 240 mL of water.
  Other Names: Olaparib
Drug: AZD5363 — Patients will be administered AZD5363 at 640 mg twice daily for two days on/five days off (2/7) schedule. Two (2) 200 mg tablets and three (3) 80 mg tablets should be taken twice daily.
  Arms: Group 2
Drug: AZD1775 — The recommended dose will be available no earlier than March 2016.
  Arms: Group 3
Drug: AZD6738 — Patients will be administered AZD6738 at 160 mg daily for days 1-7 of a 28-day cycle (7/28) schedule. AZD6738 is available as 100, 20, and 10 mg tablets. Tablets should be taken daily.
  Arms: Group 4

SUMMARY:
The primary objective of this phase II trial is to determine tumor overall response rate (ORR) in molecularly selected patients with measurable disease as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST), before versus after 16 weeks of treatment across tumor types in each arm of the study.

DETAILED DESCRIPTION:
This is a phase II signal-searching study in a range of tumor types with the potential to identify novel tumor indications for combination therapy with olaparib that can subsequently be explored in dedicated studies. Patients will be enrolled in this study based on molecular markers from genetic profiling performed on their tumors prior to study entry (outside of protocol). The trial will also identify genetic determinants of response and resistance.

Patients with tumors harboring damaging mutations in Homologous - DNA repair (HDR) genes or mutations such as ATM, CHK2, MRN (MRE11/NBS1/RAD50), CDKN2A/B and APOBEC will be treated with olaparib or olaparib and AZD6738. Enrollment to the olaparib monotherapy arm will be completed prior to commencement of enrollment to the olaparib and AZD6738 arm. Patients with tumors harboring IDH1/IDH2 mutations will be treated with olaparib. Patients with tumors harboring either TP53 or KRAS mutations or mutations in KRAS and TP53 will be treated with AZD1775 plus olaparib. Patients with tumors harboring PTEN, PIK3CA, AKT, or ARID1A mutations or other molecular aberrations leading to dysregulation of the PI3K/AKT pathway will be treated with AZD5363 plus olaparib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented metastatic cancer (solid tumors, not including hematologic malignancies)
* Patients who have received standard first-line therapy for metastatic cancer (except for the tumors for which no first-line therapy exists) and in whom a trial of targeted therapy is considered the best available treatment option. Eligible patients should not have available therapies that will convey clinical benefit.
* Progressive cancer at the time of study entry
* Measurable disease by RECIST v1.1
* Age ≥ 18 years
* Life expectancy ≥ 16 weeks
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1 (APPENDIX A: Performance Status Criteria)
* Able to understand the nature of this trial and provide written informed consent
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Molecular testing or appropriate IHC results from CLIA-certified laboratories used for patient eligibility should be obtained from the most recent tumor biopsy (baseline tumor biopsies and on-progression tumor biopsies are optional)
* No previous treatment with olaparib or any other drug sharing the same target. Prior treatment with PARP inhibitor monotherapy is allowed in the combination arms.
* Prior radiation therapy is allowed. Patients must not have received radiation therapy within 21 days prior to the initiation of study treatment.
* Other therapies: Prior experimental (non-FDA approved) therapies and immunotherapies are allowed. Patients must not have received these therapies for 21 days or five half-lives of the drug (whichever is less) prior to the initiation of study treatment and must have full recovery from any acute clinically significant effects of these therapies.
* Adequate hematologic function defined as:

  * Absolute neutrophil count (ANC) ≥ 1500/μL
  * White blood cells (WBC) > 3x109/L
  * Hemoglobin (Hgb) ≥ 10 g/dL (may be achieved with erythropoietin agents; no blood transfusions in the 28 days prior to entry)
  * Platelets ≥ 100,000/μL
  * No features suggestive of MDS/AML on peripheral blood smear
* Adequate renal and liver function defined as:

  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × the upper limit of normal (ULN) (≤ 5 × ULN if considered due to primary or metastatic liver involvement)
  * Total bilirubin ≤ 1.5 ×ULN
  * Alkaline phosphatase ≤ 2× ULN (≤ 5 × ULN if considered due to tumor)
  * Serum creatinine ≤ 1.5 ULN
* At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) or ≥ 10 mm with calipers by clinical exam OR At least one lesion (measurable and/or non-measurable) that can be accurately assessed by CT/MRI/plain x-ray/clinical exam at baseline and follow up visits.
* Women of child-bearing potential must have a negative pregnancy test (urine or serum) within 28 days prior to starting the study drug. Both males and females must agree to adequate birth control if conception is possible during the study and for 6 months after the last dose. Female patients are considered to not be of child-bearing potential if they have a history of tubal ligation or hysterectomy or are post-menopausal with a minimum of 1 year without menses.

Exclusion Criteria:

* Patients with known germline BRCA mutations in breast cancers will be excluded from the study, however testing is not required for inclusion in the study.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Prior standard of care cancer chemotherapy, immunotherapy, or radiotherapy <21 days prior to first dose of study agent(s)
* Patients with hematologic malignancies (includes patients with myelodysplastic syndrome/acute myeloid leukemia).
* Patients with primary CNS malignancies
* Patients must not have received allogeneic stem cell transplant
* Concurrent administration of any other anti-cancer therapy

  * Bisphosphonates and Denosumab for bone metastases are allowed if started at least 4 weeks prior to treatment with study agent(s).
  * Octreotide is allowed if dose is stable for >3 months with no worsening of carcinoid syndrome
  * Hormonal therapy with luteinizing hormone-releasing hormone (LHRH) analogues for medical castration in patients with castrate-resistant prostate cancer is permitted
* Patients who have not demonstrated stable recover (28 days or greater) from ≤ CTCAE grade 2 non-hematological toxicities related to prior therapy such as peripheral neuropathy or alopecia, or incomplete recovery from previous surgery, unless agreed by the Principal Investigator (PI) and documented are not eligible to participate in this study.
* Active or untreated brain metastases or spinal cord compression

  * A scan to confirm the absence of brain metastases is not required.
  * Patients with treated brain metastases or spinal cord compression are eligible if they have minimal neurologic symptoms and evidence of stable disease (for at least 1 month) or response on follow-up scan. The patient can receive a stable dose of corticosteroids before and during the study if started at least 28 days prior to initiating the study agent(s)..
* History of carcinomatous meningitis
* Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated stage I cancers (cervix, breast, colon, lung, or prostate as examples) or other advanced (> Stage I)solid tumors curatively treated with no evidence of disease for ≥ 5 years.
* Patient must not have a co-morbid condition(s) that, in the opinion of the investigator, prevent safe treatment.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV) and are receiving antiviral therapy (testing is not part of the protocol).

  - Patients with known (testing is not part of the protocol) active hepatic disease (i.e., Hepatitis B or C) due to risk of drug interactions with anti-viral therapy.
* Any of the following cardiovascular events within 6 months prior to study entry: myocardial infarction, malignant hypertension, severe/unstable angina, symptomatic congestive heart failure, cerebral vascular accident, or transient ischemic attack
* History or presence of clinically significant ventricular or atrial dysrhythmia > Grade 2 (NCI CTCAE v4.0)

  - Patients with chronic, rate-controlled atrial arrhythmias who do not have other cardiac abnormalities are eligible.
* Major surgery within 3 weeks prior to first dose of study treatment, and patients must have recovered from the effects of surgery
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g. inflammatory bowel disease) or significant bowel resection that would preclude adequate absorption
* Patients with uncontrolled seizures
* Inadequate bone marrow reserve within past 28 days prior to study treatment as demonstrated by:

  * Absolute neutrophil count (ANC) < 1500/μl,
  * WBC ≤ 3x109/L
  * Platelet count (PLT) < 100,000/μl, or
  * Hemoglobin (Hgb) < 10 g/dL
* Blood (packed red blood cells, platelets) transfusions within 1 month prior to study start
* Whole blood transfusion in the last 120 days prior to entry to the study
* Patients with concomitant use of drugs, herbal supplements and/or ingestion of foods known to strongly modulate CYP3A4 enzyme activity as specified in the drug specific appendix.
* Women who are pregnant or lactating (breastfeeding)
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Patients with a known hypersensitivity to the combination/comparator agent
* Any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results

  - Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, superior vena cava syndrome, extensive bilateral lung disease on HRCT scan or any psychiatric disorder that prohibits obtaining informed consent
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Eder, MD, Principal Investigator — Yale University Cancer Center
Locations (4):
- United States (4):
  - Yale Cancer Center, New Haven, Connecticut
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Olaparib AZD2881: Patients with cholangiocarcinoma harboring IDH 1/2 tumors will be treated with olaparib. Patients with tumors harboring mutation in HDR genes will be treated with olaparib.
  AZD2281: Patients will be administered olaparib orally twice daily (bid) at 300 mg. Two (2) x 150 mg olaparib tablets should be taken at the same times each morning and evening of each day, approximately 12 hours apart with approximately 240 mL of water.
- Olaparib & Capivasertib AZD5363: Patients with tumors harboring PTEN, PIK3CA, AKT, or ARID1A mutations or other molecular aberrations leading to dysregulation of the PI3K/AKT pathway will be treated with AZD5363 plus olaparib.
  AZD2281: Patients will be administered olaparib orally twice daily (bid) at 300 mg. Two (2) x 150 mg olaparib tablets should be taken at the same times each morning and evening of each day, approximately 12 hours apart with approximately 240 mL of water.
  AZD5363: Patients will be administered AZD5363 at 640 mg twice daily for two days on/five days off (2/7) schedule. Two (2) 200 mg tablets and three (3) 80 mg tablets should be taken twice daily.
- Olaparib & Ceralasertib AZD6738: Patients with tumors harboring either TP53 or KRAS mutations or mutations in KRAS and TP53 will be treated with AZD1775 plus olaparib. TP53 mutations must be found on the TP53 mutation eligibility list.
  AZD2281: Patients will be administered olaparib orally twice daily (bid) at 300 mg. Two (2) x 150 mg olaparib tablets should be taken at the same times each morning and evening of each day, approximately 12 hours apart with approximately 240 mL of water.
  AZD1775: The recommended dose will be available no earlier than March 2016.
- Olaparib & Adavosertib AZD1775: Patients with tumors harboring mutations in HDR genes, including ATM, CHK2, APOBEC, MRE11 complex, will be treated with AZD6738 and olaparib.
  AZD2281: Patients will be administered olaparib orally twice daily (bid) at 300 mg. Two (2) x 150 mg olaparib tablets should be taken at the same times each morning and evening of each day, approximately 12 hours apart with approximately 240 mL of water.
  AZD6738: Patients will be administered AZD6738 at 160 mg daily for days 1-7 of a 28-day cycle (7/28) schedule. AZD6738 is available as 100, 20, and 10 mg tablets. Tablets should be taken daily.
Period: Overall Study
Arm/Group | Olaparib AZD2881 | Olaparib & Capivasertib AZD5363 | Olaparib & Ceralasertib AZD6738 | Olaparib & Adavosertib AZD1775
Started | 26 | 16 | 25 | 0
Completed | 25 | 15 | 21 | 0
Not Completed | 1 | 1 | 4 | 0
Not completed — Death | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Arm 4 (Olaparib & Adavosertib AZD1775) was never activated following the study pause due to COVID.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib AZD2881 | Olaparib & Capivasertib AZD5363 | Olaparib & Ceralasertib AZD6738 | Olaparib & Adavosertib AZD1775 | Total
Number analyzed (Participants) | 26 | 16 | 25 | 0 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 11 | 19 | 0 | 47
  >=65 years | 9 | 5 | 6 | 0 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 18 | 0 | 38
  Male | 18 | 4 | 7 | 0 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 18 | 13 | 19 | 0 | 50
  Unknown or Not Reported | 8 | 3 | 5 | 0 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2
  White | 18 | 12 | 19 | 0 | 49
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 4 | 4 | 0 | 15
Region of Enrollment [Number; unit: participants]
  United States | 26 | 16 | 25 |  | 68

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Tumor overall response rate (ORR) in molecularly selected patients with measurable disease as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST), before versus after 16 weeks of treatment across tumor types in each arm of the study (Note: there will be no formal comparison between arms). Complete Response (CR): disappearance of all target lesions, Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD). Clinical Benefit is defined as the sum of CR, PR, or SD at 16 weeks from the start of treatment.
Time Frame: Change from baseline to 16 weeks
Population: 2 patients not included due to death: 1 from Olaparib AZD2881, 1 from Olaparib & Capivasertib AZD5363. The Olaparib & Adavosertib AZD1775 arm was never initiated. One participant in Olaparib & Ceralasertib AZD6738 arm not included because taken off study by physician decision and 2 subjects withdrew.
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib AZD2881 | Olaparib & Capivasertib AZD5363 | Olaparib & Ceralasertib AZD6738 | Olaparib & Adavosertib AZD1775
Number analyzed (Participants) | 25 | 15 | 24 | 0
Participants
  CR = complete response | 0 | 0 | 0 | 0
  PR = partial response | 2 | 1 | 2 | 0
  SD = stable disease | 7 | 5 | 13 | 0
  PD = progressive disease | 16 | 9 | 9 | 0

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Arm/Group | Olaparib AZD2881 | Olaparib & Capivasertib AZD5363 | Olaparib & Ceralasertib AZD6738
All-Cause Mortality (participants affected / at risk) | 1/26 | 1/16 | 0/25
Serious Adverse Events (participants affected / at risk) | 10/26 | 9/16 | 17/25
Other Adverse Events (participants affected / at risk) | 17/26 | 3/16 | 17/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib AZD2881 (N=26) | Olaparib & Capivasertib AZD5363 (N=16) | Olaparib & Ceralasertib AZD6738 (N=25)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib AZD2881 (N=26) | Olaparib & Capivasertib AZD5363 (N=16) | Olaparib & Ceralasertib AZD6738 (N=25)
Anemia (Blood and lymphatic system disorders) | 9 (21) | 2 (3) | 11 (25)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 8 (33)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (9) | 2 (4) | 8 (8)
Vomiting (Gastrointestinal disorders) | 3 (5) | 2 (3) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (4) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 0 (0) | 1 (2)
White blood cell decreased (Investigations) | 1 (2) | 0 (0) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
GGT increased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Investigations - Other (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Weight loss (Investigations) | 1 (1) | 0 (0) | 0 (0)
Fatigue (Gastrointestinal disorders) | 3 (5) | 1 (1) | 6 (7)
Fever (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (7)
Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Chills (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 3 (5)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (2)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal vascular disorder (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Immune system disorders - Other (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT02576444/Prot_SAP_000.pdf